CLINICAL TRIAL: NCT04880291
Title: A First-In-Human, Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GFB-024 as a Single Dose in Healthy Overweight and Obese Participants and as Multiple Doses in Participants With Type 2 Diabetes Mellitus
Brief Title: First-In-Human Study of GFB-024 in Healthy Overweight and Obese Participants, and Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Goldfinch Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GFB-024-102
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Kidney Diseases; Diabetic Nephropathies; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases
MeSH Terms: conditions — Kidney Diseases; Diabetic Nephropathies; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GFB-024 SAD Active (Active Comparator): Single ascending dose arm of GFB-024 treatment
  Interventions: Drug: GFB-024
- SAD Placebo (Placebo Comparator): Single ascending dose arm of placebo treatment
  Interventions: Drug: Placebo
- GFB-024 Repeat-dose Active (Active Comparator): Repeat-dose arm of GFB-024 treatment
  Interventions: Drug: GFB-024
- Repeat-dose Placebo (Placebo Comparator): Repeat-dose arm of placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFB-024 — Peripherally acting Cannabinoid-1 receptor inverse agonist monoclonal antibody
  Arms: GFB-024 Repeat-dose Active; GFB-024 SAD Active
Drug: Placebo — Matched placebo
  Arms: Repeat-dose Placebo; SAD Placebo

SUMMARY:
GFB-024 is intended for use in patients with kidney disease such as diabetic nephropathy. This study is the first time GFB-024 has been used in humans. The first part of the study will assess the safety of a single dose of GFB-024 in healthy overweight and obese volunteers and the effect of GFB-024 on the body as compared to an inactive placebo medication. The second part of the study will assess the safety of repeated doses of GFB-024 in participants with Type 2 diabetes and the effect of GFB-024 on the body as compared to an inactive placebo medication.

DETAILED DESCRIPTION:
This is a first-in-human study. It is intended to provide the initial safety, pharmacokinetics (PK), and pharmacology data for GFB-024 in humans. This study will comprise a single ascending dose (SAD) escalation component in healthy overweight and obese volunteer participants and a repeat-dose component to confirm repeat-dose safety, tolerability, PK, and immunogenicity in participants with Type 2 diabetes mellitus. It will also explore potential cannabinoid-1 receptor (CB1) activity, participant selection, pharmacodynamics, and differential response biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age at the time of signing informed consent.
* Body mass index (BMI) between 25.0 and 40.0 kg/m2, inclusive, at Screening.
* Female participants will be of non-childbearing potential.
* Male participants will agree to use contraception while on study intervention and for at least 6 months after the last dose of study intervention.
* SAD cohorts only: Participants must be in good health.
* Repeat-dose cohort only: Type 2 diabetes mellitus (T2DM) treated with lifestyle modification or metformin, and in otherwise good health except for well-controlled common conditions associated with T2DM, such as hypertension and dyslipidemia.

Exclusion Criteria:

* History of, or treatment for, psychiatric illness, including anxiety or depression within 5 years of the Screening visit.
* Participants with a history of attempted suicide or clinically significant suicidal ideation.
* History of cardiovascular disease.
* Blood pressure >155 mmHg systolic or >95 mmHg diastolic.
* History of alcoholism or drug/chemical abuse within 2 years prior to Screening.
* Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1.5 oz (45 mL) liquor, or 5 oz (150 mL) wine.
* History of significant hypersensitivity, intolerance, or allergy to more than one class of drugs.
* Positive hepatitis panel and/or positive human immunodeficiency virus test. Participants whose results are compatible with prior immunization may be included.
* SAD cohorts only: Fasting glucose >126 mg/dL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability following single ascending doses of GFB-024 | Approximately 10 weeks
  Number of participants with serious and other nonserious adverse events

SECONDARY OUTCOMES:
Safety and tolerability following repeated doses over 4 weeks of GFB-024 | Approximately 13 weeks
  Number of participants with serious and other nonserious adverse events
Characterize PK of GFB-024 following single ascending doses (Cmax) | Approximately 10 weeks
  Maximum serum concentration
Characterize PK of GFB-024 following single ascending doses (AUClast) | Approximately 10 weeks
  Area under the serum concentration-time curve from time zero to last measurable concentration
Characterize PK of GFB-024 following repeated doses (Cmax) | Approximately 13 weeks
  Maximum serum concentration
Characterize PK of GFB-024 following repeated doses (AUClast) | Approximately 13 weeks
  Area under the serum concentration-time curve from time zero to last measurable concentration
Characterize the incidence and persistence of immunogenicity of GFB-024 following single ascending doses | Approximately 10 weeks
  Number of participants with confirmed antidrug antibodies
Characterize the incidence and persistence of immunogenicity of GFB-024 following repeated doses | Approximately 13 weeks
  Number of participants with confirmed antidrug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ingela Danielsson, MD, PhD, MBA, Principal Investigator — Worldwide Clinical Trails
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No